CLINICAL TRIAL: NCT00539409
Title: Effects on Diabetic Metabolic Integrity With Treatment of Pulsatile Intravenous Insulin Therapy as Evidenced by Monitoring of Diabetic Complications.
Brief Title: Effects of Pulsatile Intravenous Insulin Therapy on Metabolic Integrity in Patients With Diabetes Mellitus
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Administrative
Sponsor: Florida Atlantic University (Other)
Collaborators: Advanced Diabetes Treatment Centers (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H09-66 Main
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, With Complications
Keywords: Diabetes Mellitus; Pulsatile Intravenous Insulin Therapy; Diabetic Quality of Life; Orthostatic Hypotension; Brittle or Labile diabetes
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus; Hypotension, Orthostatic; Diabetes Mellitus, Type 1 | interventions — Insulin; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Diabetic patients will complete quality of life questionnaires at baseline and quarterly thereafter to monitor and assess progress with complications resulting from their diabetes. Comparisons will be performed on lab values performed at baseline and every six months and medication information collected at weekly Pulsatile Intravenous Insulin treatment sessions.
- Pulsatile Intravenous Insulin Therapy (Active Comparator)
  Interventions: Procedure: Pulsatile Intravenous Insulin Therapy (Humulin R, Novolog)

INTERVENTIONS:
Procedure: Pulsatile Intravenous Insulin Therapy (Humulin R, Novolog) — Endocrinologist reviews patient activation after treatment each week and adjust the amounts of insulin and carbohydrates to be given in the next session
  Other Names: Humulin R, Novolog
  Arms: Pulsatile Intravenous Insulin Therapy

SUMMARY:
The purpose of this study is to determine if restoring normal metabolic function in patients with either type I or type II diabetes can improve the impact of the consequences of diabetic complications on the overall quality of life of diabetic patients. Patients are treated once a week with pulsatile intravenous insulin therapy mimicking normal insulin secretion. A diabetic quality of life questionnaire is completed prior to the start of the treatment and quarterly thereafter with detailed analysis performed to measure progress and outcomes

DETAILED DESCRIPTION:
It is known that the glucose metabolic pathway (glycolysis) is the primary fuel generator in the brain and nerve tissue, the heart and vascular tissue, the eye, the kidney and the liver Deficient metabolic states such as seen in the glucose metabolism of diabetics can lead to sequelae. These damaging effects are exacerbated by altered cellular metabolites, specifically the increase in catabolic and decrease in anabolic factors. It has been shown over the past twenty years that normalization of metabolism in diabetic patients can be accomplished by mimicking the normal endogenous insulin pattern (ie., in pulses). Pulsatile insulin infusion has been demonstrated to reverse the diabetic metabolic state from primary fat utilization to carbohydrate utilization. This has been correlated with a stabilization of kidney function in patients with overt diabetic nephropathy, stabilization of blood glucoses, stabilization of blood pressure patterns, and reversal of hypoglycemic unawareness.

The Diabetes Quality Of Life questionnaire was developed to assess quality of life in patients with types 1 and 2 Diabetes Mellitus. This study measures whether the reversal of abnormal metabolism in patients with diabetes is correlated with an improvement in their quality of life.The respiratory quotient (RQ) is a measurement of CO2 exhaled and O2 inhaled and is proportionate to the fuel sources being used by the body, primarily the liver over short periods of time. The higher the RQ, the more glucose and less alternative fuel sources are being utilized. Following the RQ change helps determine the effectiveness of physiological insulin administration in increasing anabolic functions in diabetic individuals. By improving the body's glucose metabolism and thereby causing beneficial effects of anabolic factors, the possibility of serious complications can be decreased. In addition the use of oral carbohydrate at the same time along with the physiologic insulin administration stimulates the appropriate gut hormones which augment this effect, a response which cannot be duplicated with intravenous glucose. The purpose of our studies is to determine whether the physiologic administration of insulin along with the augmenting effect of oral carbohydrates will normalize metabolism in diabetic patients and improve their quality of life indices.

The RQ is determined by the use of a metabolic cart. Individuals breathe into a mask for 3-5 minutes after a rest period of 30 or more minutes. The ratio of exhaled volume of CO2 to the inhaled volume of O2 is determined as the RQ. The physiologic range is 0.7 to1.3. Individuals using fat as a primary fuel have a ratio of 0.7, protein or mixed fuels is 0.8-0.9 and carbohydrate is 0.9-1.0. Those taking excessive calories will have RQ's higher than 1.05. The RQ can be followed serially and this is done before and after each pulsatile IV insulin treatment, during the 3 successive sessions on a single treatment day. The amount of intravenous insulin and oral glucose given is determined by the RQ changes during the previous session.pulsatile IV insulin therapy encourages the glucose metabolism in diabetics to normalize in multiple organs, especially muscle, retina, liver, kidney and nerve endings. The process fundamentally requires the administration of high dose insulin pulses similar to those found in non diabetic humans by their pancreas into the surrounding portal circulation. Oral carbohydrates are given simultaneously to augment the process and prevent hypoglycemia. The process is monitored by frequent glucose levels and respiratory quotients (RQ). RQ is measured by a metabolic cart which determines the ratio VCO2/ VO2. This ratio is specific for the fuel used at any one time by the body. The glucose levels are monitored to keep glucose levels appropriate and the RQ determines the need to readjust the infusion protocol in each patient for subsequent insulin infusion sessions.Patient is evaluated post session and discharged when stable.

Frequent monitoring of RQ is necessary as these levels change rapidly, depending on the fuel being utilized by the body. Pulsatile IV insulin therapy shifts metabolism from primarily fatty acid metabolism to primarily glucose metabolism. This shift is reflected by the increase in respiratory quotient. However during rest periods the RQ may fall back to lower levels. Therefore RQ's are done at the beginning and at the end of each insulin infusion session of 1 hour in order to appropriately monitor and adjust insulin and carbohydrate loads to reach optimal activation in each session.

ELIGIBILITY:
Inclusion Criteria:

* The researchers will include up to 750 pts between male and female between -the ages of 21 and 85 diagnosed with diabetes mellitus
* Self reporting or diagnosed with significant complications resulting from diabetes
* Taking oral agents and/or insulin for diabetic control
* Under an Endocrinologist supervision for their diabetes management, Endocrinologist must assess and approve pt for participation in this study
* Ability to swallow without difficulty
* Ability to perform Respiratory Quotient requirements by breathing into a mask for 3 minutes at a time

Exclusion Criteria:

* Lack of Intravenous access
* Pregnancy
* Alcohol abuse, drug addiction or the use of illegal drugs
* Active liver disease
* Active chemotherapy
* Positive HIV
* Inability to breathe into a respiratory quotient machine

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2006-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Monitor and assess whether Pulsatile Intravenous Insulin Therapy can effect Metabolic Integrity in patients with Diabetes Mellitus. Monitor results of QOL questionnaires, Hgb A1C levels, medications to see if patients complications improve | Diabetes Quality of Life questionnaires are completed at baseline and every quarter thereafter, Lab values are collected at baseline and every 6 months thereafter, current medications are collected weekly

CONTACTS AND LOCATIONS:
Overall Officials: Betty Tuller, PhD, Principal Investigator — Florida Atlantic University
Locations (1):
- Florida Atlantic University, Boca Raton, Florida, United States